CLINICAL TRIAL: NCT05334290
Title: Financial Toxicity and Patient-Reported Outcomes in Italian Patients Affected by Gastroenteropancreatic Neuroendocrine Neoplasms (GEP-NEN)
Brief Title: Financial Toxicity and Patient-Reported Outcomes in GEP-NEN During Treatment
Acronym: FiReNEN
Status: Recruiting | Type: Observational
Sponsor: Massimo Falconi (Other)
Responsible Party: Sponsor-Investigator, Massimo Falconi, Head od Pancreatic Surgery Unit, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Other Study IDs: FiReNEN
Record Dates: First submitted 2022-03-30; First posted 2022-04-19 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Neuroendocrine Tumors
Keywords: GEP-NEN; financial toxicity; Quality of life; Costs
MeSH Terms: conditions — Neuroendocrine Tumors; Financial Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate the financial toxicity reported by Italian patients affected by GEP-NEN during the first year of treatment after diagnosis and its correlations with patient-reported outcomes (PROs) and quality of life (QoL).

DETAILED DESCRIPTION:
Gastroenteropancreatic neuroendocrine neoplasms (GEP-NEN) are rare tumours whose incidence has increased during the years. However, referral centers specialized in diagnosis and treatment of these diseases are few. So, patients may be forced to travel long distances in order to reach a disease specialized center (ENETS certification) to plan the correct management and receive the better treatment. On the other hand, patients could research different clinical consulting by several medical specialists without clear indication. Moreover, today also advanced disease allows the patients a good prognosis with long survival. The resulting emotional and psychological burden may contribute to the worse quality of life. Therefore, patients with GEP-NEN have a deal with the financial consequences related to the diagnosis and treatment of their disease including out of pocket costs, loss of income and caregiver burden. Financial toxicity, defined as subjective financial concerns of cancer and objective financial consequences, has been investigated in this study in Italian patients affected by GEP-NEN

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* New diagnosis of gastroenteropancreatic neuroendocrine neoplasms (GEP-NEN)
* Patients who are candidates for surgical and/or medical treatment [including somatostatin analogues (SAA), peptide recector radionuclide therapy (PRRT), target therapies (everolimus or sunitinib) and chemotherapy];
* Signed informed consent

Exclusion Criteria:

* Age < 18 years
* Patients diagnosed with GEP-NEN who are candidates for a surveillance management.
* Patients diagnosed with GEP-NEN who are candidates for best supportive care and/or have a life expectancy < 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls individuals (>18 years) with a new diagnosis of GEP-NEN who are candidates for surgical and/or medical treatment, in Italian Centers. Are excluded from this study patients candidates for a surveillance management and, on the opposite side, with life expectancy < 6 months or candidates for best supportive care.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-08-06 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2024-08-05 (Estimated)

PRIMARY OUTCOMES:
Financial toxicity | 12 months
  Financial toxicity measured by Comprehensive Score for financial toxicity (COST) and out of pockets.
Quality of Life (QoL) | 12 months
  Evaluate the QoL of patients affected by GEP-NEN, as measured by the Questionnaires assessing the QoL of Cancer Patients (QLQ-C30)

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Partelli, Professor, Principal Investigator — San Raffaele Hospital Milan
Locations (1):
- IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Singh S, Granberg D, Wolin E, Warner R, Sissons M, Kolarova T, Goldstein G, Pavel M, Oberg K, Leyden J. Patient-Reported Burden of a Neuroendocrine Tumor (NET) Diagnosis: Results From the First Global Survey of Patients With NETs. J Glob Oncol. 2016 Jun 8;3(1):43-53. doi: 10.1200/JGO.2015.002980. eCollection 2017 Feb. PMID 28717741
- [Result] de Souza JA, Yap BJ, Wroblewski K, Blinder V, Araujo FS, Hlubocky FJ, Nicholas LH, O'Connor JM, Brockstein B, Ratain MJ, Daugherty CK, Cella D. Measuring financial toxicity as a clinically relevant patient-reported outcome: The validation of the COmprehensive Score for financial Toxicity (COST). Cancer. 2017 Feb 1;123(3):476-484. doi: 10.1002/cncr.30369. Epub 2016 Oct 7. PMID 27716900
- [Result] Beaumont JL, Cella D, Phan AT, Choi S, Liu Z, Yao JC. Comparison of health-related quality of life in patients with neuroendocrine tumors with quality of life in the general US population. Pancreas. 2012 Apr;41(3):461-6. doi: 10.1097/MPA.0b013e3182328045. PMID 22422138